CLINICAL TRIAL: NCT06245785
Title: Liver Resection for Patients With Hepatocellular Carcinoma and Impaired Liver Function: A Chinese Multicenter Observational Study
Brief Title: Liver Resection for Patients With Hepatocellular Carcinoma and Impaired Liver Function
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: liu lei
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Hepatic Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- liver resection
- transarterial chemoembolisation
  Interventions: Procedure: transarterial chemoembolisation

INTERVENTIONS:
Procedure: transarterial chemoembolisation — Before TACE, hepatic arteriography was performed to evaluate the vascular anatomy and tumour vascularity. During TACE, a vascular catheter was selectively inserted into the tumour-feeding artery with an injection containing a mixture of doxorubicin (10-50 mg) and lipiodol (2-20 mL), followed by embolisation using gelatin sponge particles. TACE was repeated when residual viable tumours were confirmed or new lesions developed in patients with adequate liver function. Laboratory assessments were performed every four to six weeks. Radiological evaluation using contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) was recommended during weeks 4 and 8 after treatment and every 8 weeks thereafter. However, in clinical practice, the intensity of follow-up depends on an individual's baseline characteristics and response to the last treatment.
  Groups: transarterial chemoembolisation

SUMMARY:
Hepatic dysfunction limits the therapeutic options for hepatocellular carcinoma (HCC), which is closely associated with patient prognosis. Established practice guidelines for patients with HCC and impaired liver function are lacking. The treatment allocation in these populations is heterogeneous and remains controversial. This study compared the survival benefits of liver resection (LR) and transarterial chemoembolisation (TACE) in patients with HCC and impaired liver function.

ELIGIBILITY:
Inclusion Criteria:

* patients with HCC who received conventional LR or TACE

Exclusion Criteria:

* （1） presence of portal vein tumour thrombosis (PVTT), hepatic artery, biliary duct or inferior vena cava invasion
* （2） extrahepatic spread (EHS)
* （3） albumin-bilirubin grade 1 or 3
* （4） Eastern Cooperative Oncology Group Performance Status (ECOG-PS) >1
* （5） tumour number >3
* （6） other tumours or severe cardiac, cerebral, and renal insufficiency
* （7）ascites, hepatic encephalopathy, and jaundice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study data were extracted from a nationwide database of patients with HCC treated at 15 Chinese centres between January 2012 and December 2022.We included patients who were diagnosed with HCC according to the American Association for the Study of the Liver Disease/European Association for the Study of the Liver Guidelines and who received conventional LR or TACE
Sampling Method: Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 year
  The overall survival rate at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: zhao s jie, Principal Investigator — Teachers and students
Locations (2):
- China (2):
  - Tangdu hospital, Xi'an, Shaanxi
  - Xijing hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No